CLINICAL TRIAL: NCT03345290
Title: Impact of the Central Blood Pressure Level in Cerebral Metabolic Aging: a 18F-FDG PET Study.
Acronym: PACTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, MD, PhD, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PSS2016/PACTEP-VERGER/VS
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Aging Disorder
Keywords: Aging; Central pressure; FDG PET
MeSH Terms: interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects (Experimental): Subjects referred to a FDG PET scan (standard PET without cerebral step) without any oncologic setting. Patients will be included as following critera: 25% of subjects will have under 40 years old, 25% between 40 and 60 yeard old et 50% higher than 60 years old.
  Interventions: Device: PET with a cerebral step; Device: Central blood pressure measurement; Other: Neurocognitive tests

INTERVENTIONS:
Device: PET with a cerebral step — Positron Emission Tomography with a cerebral step before to carry out the standard Position Emission Tomography
Device: Central blood pressure measurement — Central blood pressure measurement
Other: Neurocognitive tests — Mini Mental State Examination, MMSE, Mini International Neuropsychiatric Interview MINI and Frontal Assessment Batery FAB

SUMMARY:
Cerebral glycolytic metabolism can be quantified by quantitative analysis of 18F-Fluorodeoxyglucose (18F-FDG) Positron Emission Tomography (PET). This allows to identify neurological diseases at an early stage of functional abnormalities, before any anatomical lesions, and to differentiate them from the "normal" brain aging. Aging mainly leads to atrophy with a decrease in cerebral metabolism in the prefrontal cortex, with consequent deterioration of cognitive processes, in particular executive functions (5).

In a population of 92 "control" subjects, investigators have already quantified the importance of the aging in frontal cortex hypometabolism. These patients were referred for a 18F-FDG PET in the follow-up of lymphoma considered to be in complete remission (PET without cerebral step), without any chemoradiotherapy within 2 months and with normal neuropsychological tests (Mini Mental State Examination, MMSE, Mini International Neuropsychiatric Interview MINI and Frontal Assessment Battery FAB).

However, cerebral aging can be "accelerated" by vascular risk factors, including increased central blood pressure, as investigators have recently reported in a pilot study involving elderly patients. This central pressure, which is directly linked to the cerebral micro-vascularization, can be easily measured by applanation tonometry. In this pilot study, investigators showed that a central pulse pressure equal or greater than 50 mmHg was associated with a significant frontal hypometabolism in elderly patients. This confirmed, at a stage of pre-clinical remodeling, the worse prognostic significance for this criterion, as reported in large epidemiological studies (increased risk of stroke and cardiac vascular events).

However, it is not yet known whether the level of central blood pressure interfere with the brain metabolism of younger subjects, especially with regard to aging observed throughout life. If this hypothesis is confirmed, preventive therapeutic strategies for accelerated aging, could thus integrate the monitoring of central pressure and cerebral metabolism.

The objective of this study is to determine, in a population of control subjects and on a larger scale, the impact of central blood pressure on brain metabolic aging , by using 18F-FDG PET.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old, with written informed consent,
* Subjects referred for 18F-FDG PET in a non-oncological setting,
* Absence of pregnancy or breastfeeding,
* Lack of chemotherapy in the previous year and no cerebral radiotherapy.
* No history of psychiatric or neurological pathology.
* Absence of treatment with psychotropic action, and absence of corticosteroids.

Exclusion Criteria:

* "abnormal" neuropsychological tests:

  * Mini Mental State Examination (MMSE) <27,
  * Current major depressive episode on the Mini International Neuropsychologic Interview (MINI),
  * Frontal Assessment Battery (FAB) <15.
* 18F-FDG PET examination showing ischemic, neurodegenerative, neoplastic or other brain lesions (independent of a normal or accelerated aging process).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
volume of brain areas detected by quantitative analysis | At inclusion
topography of brain areas detected by quantitative analysis | At inclusion
central blood pressure | At inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Verger, MD, PhD, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hurstel M, Joly L, Imbert L, Zimmermann G, Roch V, Schoepfer P, Lamiral Z, Salvi P, Benetos A, Verger A, Marie PY. Volume of the proximal half of the thoracic aorta is the most comprehensive FDG-PET/CT indicator of arterial aging throughout adulthood. Eur J Hybrid Imaging. 2023 Jun 28;7(1):11. doi: 10.1186/s41824-023-00169-2. PMID 37369917